CLINICAL TRIAL: NCT00923871
Title: Automating the Breast Radiation Therapy Process to Improve Efficiency
Brief Title: Automating Breast Radiation Therapy (RT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 09-0197-CE
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: CBCT; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cone Beam CT (Experimental)
  Interventions: Procedure: Cone Beam CT

INTERVENTIONS:
Procedure: Cone Beam CT — Patients will also have a CBCT scan when they are having their first IMRT treatment.

SUMMARY:
Breast radiation treatment is planned from a Computed Tomography (CT) scan. This study is designed to investigate a method to reduce the time between the planning of radiation treatment and its actual start by automating the intensity-modulated radiation therapy (IMRT) planning process. The investigators plan to examine data from another scan called Cone Beam Computed Tomography (CBCT). A CBCT scan provides similar information to a conventional CT scan, however the images for CBCT are acquired at the treatment unit (linear accelerator used for treatment). Using these x-ray pictures of patients, the study team consisting of a radiation oncologist, a medical physicist and a radiation therapist will create a custom treatment plan unique to each patient. By doing this, the investigators hope to reduce the amount of time spent waiting for treatment and the number of hospital visits for patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer who will receive standard two-field tangential whole breast radiation therapy with dose prescription of 4240 cGy in 16 fractions, 5000 cGy in 25 fractions or 4000 cGy in 16 fractions.
* Patients with any stage of breast cancer.
* Patients with prior treatment such as surgery or chemotherapy for any type of cancer.
* Able to provide a written informed consent.
* 18 years of age or older.

Exclusion Criteria:

* < 18 years of age.
* Unable to provide informed consent.
* Males.
* Patients who received partial breast radiation and not the standard dose.
* Patients who will not receive 4240 cGy in 16 fractions, 5000 cGy in 25 fractions, or 4000 cGy in 16 fractions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-06; Primary Completion 2015-01-05 (Actual); Study Completion 2016-04-29 (Actual)

PRIMARY OUTCOMES:
To generate on-line IMRT treatment plans using automated tools based on CBCT images acquired at the treatment unit. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Koch, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada